CLINICAL TRIAL: NCT04764188
Title: A Multicenter Non-Interventional Cohort Study to Evaluate the Real-World Clinical Management and Outcomes of Patients Diagnosed With ALK-Positive Advanced NSCLC Treated With Alectinib (ReAlec)
Brief Title: An Observational Study to Evaluate the Real-World Clinical Management and Outcomes of ALK-Positive Advanced NSCLC Participants Treated With Alectinib
Acronym: ReAlec
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO42122
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
Keywords: ALK-positive NSCLC
MeSH Terms: interventions — alectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Participants starting alectinib treatment after (Arm A) or before (Arm B) study enrollment as first-line treatment will be followed up for up to 4 years.
  Interventions: Drug: Alectinib
- Cohort 2: Participants receiving alectinib as second-line treatment after study enrollment will be followed up for up to 2 years.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive alectinib in accordance with local clinical practice and local labeling.

SUMMARY:
This study aims to characterize the clinical management and outcomes of participants diagnosed with anaplastic lymphoma kinase (ALK)-positive advanced non-small cell lung cancer (NSCLC) who are being treated with alectinib in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of advanced NSCLC (stage IIIB, IIIC, IVA, or IVB) on or after the date of local approval for alectinib as first-line treatment and/or second-line treatment for ALK-positive advanced NSCLC and planned to receive treatment as per routine for at least one cycle (28 days) while on study
* ALK-positive as confirmed by immunohistochemistry (IHC), fluorescent in situ hybridization (FISH), next generation sequencing (NGS), or other non-specified sequencing methods, documented prior to receiving treatment with an ALK inhibitor
* Cohort 1: Currently receiving, or planned to receive, treatment for ALK-positive advanced NSCLC with alectinib as first-line treatment
* Cohort 2: Planned to receive treatment for ALK-positive advanced NSCLC with alectinib as second-line treatment
* Able to be followed-up by participating site
* Participants with advanced NSCLC who have CNS metastases are eligible for inclusion

Exclusion Criteria

* Participants not receiving alectinib for the treatment of ALK-positive advanced NSCLC according to standard of care and in line with local product information
* Participants not receiving the Roche studied medicinal product
* Participants who have received or are currently receiving alectinib as an investigational study drug in a clinical trial for the treatment of advanced NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be identified in real-world clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Investigator-Confirmed Progression-Free Survival (PFS) According to the Local Standard of Care or per Response Evaluation in Solid Tumors (RECIST) - Cohort 1 | From the first administration of alectinib to the date of first documentation of disease progression, or death due to any cause, whichever occurs first (up to 4 years)
Investigator-Confirmed PFS According to the Local Standard of Care or per RECIST - Cohort 2 | From the first administration of alectinib to the date of first documentation of disease progression, or death due to any cause, whichever occurs first (up to 2 years)
Choice of the Next Line of Treatment (LoT) Post-Alectinib | Up to approximately 1 year
Duration of Next LoT | Up to approximately 1 year
Reasons for Discontinuation of Next LoT | Up to approximately 1 year

SECONDARY OUTCOMES:
Time to Loss of Clinical Benefit (TTLCB) | From the first administration of alectinib to loss of clinical benefit as assessed by the treating physician (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Overall Survival (OS) | From the first administration of alectinib to death from any cause (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Objective Response Rate (ORR), Defined as a Complete Response (CR) or Partial Response (PR) | From the first administration of alectinib to first CR or PR (up to 4 years for Cohort 1 and Cohort 2)
Time to Response | From the first administration of alectinib to first CR or PR (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Duration of Objective Response (DOR) | From first documentation of CR or PR (whichever occurs first) after the first administration of alectinib until death or progressive disease (PD) (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Disease Control Rate (DCR) | At least 12 weeks after the first administration of alectinib (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Duration of Disease Control | Time from the first administration of alectinib to the first documentation of CR, PR, or stable disease (whichever occurs first), until death or PD (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Time to Central Nervous System (CNS) Progression (Cohort 1 Arm A) | Time interval from the first administration of alectinib to the date of confirmed CNS metastases in participants with no CNS metastases at baseline (up to 4 years)
Time to Initiation of Next Line of Treatment (LoT) | From the first administration of alectinib to the date of initiation of next LoT or death due to any cause, whichever occurs first (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Quality of Life Status Using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scores | At enrollment and every 3 months thereafter (up to 4 years for Cohort 1 and 2 years for Cohort 2)
Quality of Life Status Using the EORTC QLQ-LC13 Scores (Cohort 1 Arm A and Cohort 2) | At enrollment and every 3 months thereafter (up to 4 years for Cohort 1 and 2 years for Cohort 2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (116):
- Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires, Argentina
- Australia (6):
  - Lifehouse, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter MacCallum Cancer Center, East Melbourne, Victoria
- Austria (3):
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
  - Klinik Penzing, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (7):
  - CHIREC, Auderghem
  - AZ Sint Lucas (Sint Lucas), Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - CHU de Liège, Liège
  - AZ Glorieux- vzw Werken Glorieux, Ronse
  - Vitaz, Sint-Niklaas
- Bulgaria (5):
  - Complex Oncology Center Burgas, Burgas
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
  - DDODIU-Plovdiv, EOOD, Plovdiv
  - MBAL Serdika EOOD, Sofia
  - Acibadem City Clinic Tokuda, Sofia
- Chile (2):
  - Inst. Nacional Del Torax, Santiago, Santiago Metropolitan
  - Centro de Estudios Clínicos SAGA, Santiago
- China (14):
  - Hu Nan Provincial Cancer Hospital, Changsha
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangzhou Panyu Central Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Anhui Chest Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Cancer Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center, Wuhan
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
- Colombia (4):
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Hospital Universitario San Ignacio, Bogotá
  - Angiografia del Occidente, Cali
  - Instituto Cancerología Medellin, Medellín
- Croatia (2):
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Centre Zagreb, Zagreb
- Cuba (2):
  - Hospital Hermanos Ameijeiras, La Habana
  - Instituto Nacional de Oncología y Radiología (INOR), La Habana
- Czechia (3):
  - Masaryk?v onkologický ústav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Thomayerova nemocnice, Praha 4 - Krc
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Ichilov Sourasky Medical Center, Tel Aviv
- Italy (16):
  - Presidio Ospedaliero Centrale, Taranto, Apulia
  - Grande Ospedale Metropolitano, Reggio Calabria, Calabria
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Fondazione Ptv Policlinico Tor Vergata, Rome, Lazio
  - Policlinico Universitario "Agostino Gemelli", Rome, Lazio
  - AZ. Ospedaliera San Giovanni - Addolorata, Rome, Lazio
  - A.O. Villa Scassi, Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Asst Di Cremona, Cremona, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Ospedale Oncologico A.Businco, Cagliari, Sardinia
  - AO Ospedali Riuniti Villa Sofia-Cervello-Presidio Ospedaliero Cervello, Palermo, Sicily
  - Ospedale San Jacopo, Pistoia, Tuscany
  - Clinica Oncologica-Ospedali Riuniti Ancona, Torrette, Tuscany
  - Ospedale Silvestrini, Perugia, Umbria
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Public Institution, Kaunas
  - National Cancer Institute, Vilnius
- Instituto Oncológico Nacional (ION), Panama City, Panama
- Peru (3):
  - Aliada Centro Oncologico, Lima
  - Oncosalud Sac, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
- Portugal (2):
  - Hospital de Sao Joao, Porto
  - CHVNG/E_Unidade 1, Vila Nova de Gaia
- Romania (7):
  - Alba Emergency County Hospital, Alba Iulia
  - Emergency University Bucharest Hospital, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Amethyst Cluj, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - Centrul de Oncologie Oncohelp, Timișoara
- Russia (5):
  - Altai Regional Oncological Center, Barnaul, Altayskiy Kray
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky, Krasnoyarsk, Krasnodarskiy Kray
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk, Moscow Oblast
  - LLC "Oncology scientific centre", Pesochny, Sankt-Peterburg
- Serbia (4):
  - Clinic for Pulmonology, Clinical Center of Serbia, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
  - Clinical Center Nis, Niš
- Turkey (Türkiye) (15):
  - Adana Baskent University Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Ataturk Sanatoryum Egitim Ve Arastirma Hastanesi, Ankara
  - Gazi University Medical Faculty, Oncology Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara City Hospital, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Pamukkale University School Of Medicine, Denizli
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital, Istanbul
  - Izmir Dr. Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Inonu University Medical Faculty of Medicine, Malatya
  - Necmettin Erbakan Üniversitesi Meram T?p Fakültesi Yunus Emre, Meram
- United Arab Emirates (2):
  - Mediclinic Airport Road Hospital, Abu Dhabi
  - Mediclinic City Hospital, Dubai
- Sanatorio CASMU, Montevideo, Uruguay
- Vietnam (3):
  - Hanoi Oncology Hospital, Hanoi
  - K hospital, Hanoi
  - Hochiminh city oncology hospital, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing